CLINICAL TRIAL: NCT00556621
Title: Phase 1-2 Study of the Association of Gemzar ® - Cisplatin-concurrent Radiotherapy in Patients With Non-metastatic Tumors of the Bladder
Brief Title: Gemcitabine, Cisplatin, and Radiation Therapy in Treating Patients With Stage II or Stage III Bladder Cancer
Acronym: GEMCIRAV
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Collaborators: Groupe D'Etude des Tumeurs Uro-Genitales (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000574107; CLCC_GEMCIRAV; INCA-RECF0285; GETUG-CLCC-GEMCIRAV
Record Dates: First submitted 2007-11-09; First posted 2007-11-12 (Estimated); Last update posted 2015-07-30 (Estimated); Status verified 2015-07

CONDITIONS: Bladder Cancer
Keywords: stage II bladder cancer; stage III bladder cancer; transitional cell carcinoma of the bladder
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Cisplatin; Gemcitabine; Biopsy; Cystoscopy; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- gemcitabine, cisplatine, radiotherapy (Other)
  Interventions: Drug: cisplatin; Drug: gemcitabine hydrochloride; Procedure: biopsy; Procedure: cystoscopy; Procedure: therapeutic conventional surgery; Radiation: radiation therapy

INTERVENTIONS:
Drug: cisplatin
Drug: gemcitabine hydrochloride
Procedure: biopsy
Procedure: cystoscopy
Procedure: therapeutic conventional surgery
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as gemcitabine and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving combination chemotherapy together with radiation therapy may kill more tumor cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of gemcitabine when given together with cisplatin and radiation therapy and to see how well they work in treating patients with stage II or stage III bladder cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the incidence and nature of acute and late toxicity of gemcitabine hydrochloride, cisplatin, and concurrent radiotherapy in patients with stage II or III transitional cell carcinoma of the bladder. (Phase I)
* Determine the efficacy of this regimen, in terms of local tumor control (absence of local progression), in these patients. (Phase II)

Secondary

* Determine the maximum tolerated dose and the recommended phase II dose of gemcitabine hydrochloride when administered with cisplatin and radiotherapy in these patients. (Phase I)
* Assess the 5- and 10-year survival and the progression-free survival of patients treated with this regimen. (Phase II)
* Assess the quality of life of patients treated with this regimen. (Phase II)

OUTLINE: This is a phase I, dose-escalation study of gemcitabine hydrochloride followed by a phase II, multicenter study.

Patients receive gemcitabine hydrochloride IV over 30 minutes twice weekly for 5 weeks and cisplatin IV continuously over 4 days on days 2-5 and 23-26 (weeks 1 and 4). Patients also undergo radiotherapy once daily 5 days a week for 5 weeks.

Three weeks after completion of treatment, patients undergo cystoscopy and transurethral resection (TUR). Patients with residual tumor or disease progression undergo radical TUR. After surgery, patients who achieve a complete response receive gemcitabine hydrochloride IV twice weekly for 2 weeks and cisplatin IV continuously over 4 days in week 1. Patients also undergo radiotherapy once daily 5 days a week for 2 weeks.

After completion of study treatment, patients are followed at 6-8 weeks and then 6 months thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of muscle invasive transitional cell carcinoma of the bladder

  * T2-4a, N0, M0 (stage II or III disease)
* No adenocarcinoma or squamous cell carcinoma

PATIENT CHARACTERISTICS:

* WHO performance status (PS) 0-2 or Karnofsky PS 70-100%
* Life expectancy ≥ 6 months
* ANC ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 10 g/dL
* Creatinine clearance ≥ 60 mL/min
* Not pregnant or nursing
* Fertile patients must use effective contraception during and for at least 2 months after completion of study treatment
* No other prior malignancy, except previously treated nonmalignant skin cancer or carcinoma in situ of the cervix
* No prior serious digestive complications (e.g., ulcerative colitis or complicated diverticulosis)

PRIOR CONCURRENT THERAPY:

* No prior radiotherapy or chemotherapy (except for intravesical instillations)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2005-06; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Incidence and nature of acute and late toxicity (Phase I) | From baseline to the end of treatment
Local tumor control (Phase II) | From baseline to the end of treatment

SECONDARY OUTCOMES:
Maximum tolerated dose and recommended phase II dose of gemcitabine hydrochloride when administered with cisplatin and radiotherapy (Phase I) | From baseline to the end of treatment
5- and 10-year survival (Phase II) | until 5 and 10 year after the end of treatment
Progression-free survival (Phase II) | 6 to 8 weeks after to the end of treatment
Quality of life (Phase II) | From baselin to the end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: David Azria, MD, PhD, Study Chair — Institut du Cancer de Montpellier - Val d'Aurelle
Locations (1):
- Centre Regional de Lutte Contre le Cancer - Centre Val d'Aurelle, Montpellier, France